CLINICAL TRIAL: NCT03269422
Title: A Phase I Feasibility Study of Radiotherapy to the Prostate and Dominant Intra-Prostatic Lesion (DIL) Using Ultra-Hypofractionated, MR Image-Guided, Intensity-Modulated Radiotherapy
Brief Title: Radiotherapy to the Prostate and Dominant Intra-Prostatic Lesion (DIL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-407
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: 17-407; Intermediate Risk Prostate Cancer; DIL; Dominant Intra-Prostatic Lesion
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MR Image Guided, Intensity-Modulated Radiotherapy (Experimental): Patients enrolled in this study will undergo MR-based, image-guided, intensity-modulated radiotherapy using similar equipment, techniques, and treatment-planning procedures as currently practiced at MSKCC.
  Interventions: Radiation: MR-based image-guided, intensity-modulated radiotherapy

INTERVENTIONS:
Radiation: MR-based image-guided, intensity-modulated radiotherapy — Patients will receive a standard dose of 8 Gy/fraction for five fractions for a total dose of 40 Gy to the prostate with a simultaneously delivered boost of 9 Gy for five fractions (clinically non-standard dose of 45 Gy total) to a single dominant lesion with a maximum dimension of at least 0.5 cm as determined on pre-treatment diagnostic T2 MRI imaging.

SUMMARY:
The purpose of the study is to find out the feasibility and effects of ultra-hypofractionated radiotherapy to the prostate and dominant lesion as definitive treatment for intermediate risk prostrate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate risk prostate cancer patients will be eligible for this study. Risk groups will be assigned as per NCCN guidelines. Intermediate risk patients will be defined as:

  * PSA 10-20 ng/ml or
  * Gleason score = 7 or
  * Clinical stage T2b/T2c
* Additionally, patients will be required to meet the following criteria:

  * Age >18
  * KPS > 80
  * Prostate size < 60cc
  * Presence of a prostatic lesion with maximum dimension of >/= 0.5cm and no more than two additional disease foci, each with a maximum dimension less than that of the dominant lesion.
  * International Prostrate Symptom Score < 15
  * Subjects must fill out the standard MRI screening form and satisfy all MRI screening criteria

Exclusion Criteria:

* Prior androgen deprivation therapy for prostate cancer
* Evidence of metastatic disease on bone scan or MRI/CT
* MRI ineligibility due to the presence of a cardiac pacemaker, defibrillator or other implanted metallic or electronic device which is considered MR unsafe, severe claustrophobia or inability to lie flat for the duration of the study, etc.
* Metallic hip implant, metallic implant or device in the pelvis that might distort the local magnetic field and compromise quality of MP-MRI.
* Lateral pelvic separation greater than 50 cm and/or anterior-posterior separation greater than 35 cm which are incompatible with MRCAT reconstruction
* Contra-indications to receiving gadolinium contrast
* KPS < 80
* Pelvic MRI or CT (MRI preferred) evidence of radiographic T3, T4 or N1 disease.
* Prior history of transurethral resection of the prostate
* Prior history of chronic prostatitis
* Prior history of urethral stricture
* Prior history of pelvic irradiation
* History of inflammatory bowel disease
* Unable to give informed consent
* Unable to complete quality of life questionnaires
* Abnormal complete blood count. Any of the following

  * Platelet count less than 75,000/ml
  * Hb level less than 10 gm/dl
  * WBC less than 3.5/ml
* Abnormal renal function tests (creatinine > 1.5)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Treatment related toxicity of ultra-hypofractionated radiotherapy will be assessed according to NCI CTCAE v3.0 gastrointestinal or genitourinary toxicity | 36 months
  Assess toxicity of ultra-hypofractionated radiotherapy to the prostate and dominant lesion as definitive treatment for intermediate risk prostate cancer. Severe Toxicity will be assessed and defined as Grade 3 or higher NCI CTCAE v3.0 gastrointestinal or genitourinary toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gorovets, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only and follow up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and follow up), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org